CLINICAL TRIAL: NCT00715325
Title: Evaluation of Safety and Efficacy of a New Colonoscope, ProtectiScope CS, to Diagnose Large Bowel Diseases
Brief Title: ProtectiScope CS Intended for Diagnostic and Therapeutic Colonoscopy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stryker GI Ltd. (Industry)
Responsible Party: Dr. Ori Segol, Carmel Nedical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CSP-IL-LIT-0703_S_01
Record Dates: First submitted 2008-07-13; First posted 2008-07-15 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Colon Cancer
Keywords: colonoscopy; disposable; single use
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Device: Protectiscop CS

INTERVENTIONS:
Device: Protectiscop CS — Patients who are indicated for screening colonoscopy will be recruited into the trial. The ProtectiScope CS sleeve is assembled on the colonoscope.standard colonoscopy is performed. Subjects will be followed for 1-month post procedure.

SUMMARY:
The purpose of this study is to determine whether the ProtectiScope CS is capable to perform diagnostic and therapeutic colonoscopy.

DETAILED DESCRIPTION:
The ProtectiScope CS is a disposable-based colonoscope incorporating a miniature video camera,integral light source along with single-use sleeves and application Channels.

The ProtectiScope CS is intended to provide visualization and therapeutic access to the Lower Gastrointestinal Tract, in adult patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Subject between the ages of 18 and 80
* Subject is indicated for screening colonoscopy
* Subject is willing to sign informed consent form

Exclusion Criteria:

* Subject is suspected, based on radiographic or other clinical grounds, of suffering from one or more of the following: full or partial colonic obstruction; acute abdomen; gross hematochezia; severely ulcerated colon; diverticulitis; severe diverticulosis; toxic megacolon.
* Subject has active cardiac problems and history of heart failure, severe pulmonary diseases renal failure (creatinine >2) uncontrolled diabetes and any other illness judged by investigator to substantiate exclusion.
* Subject has a history of significant other diseases.
* Subject has a history of psychiatric disorders which would prevent compliance with study instructions
* For female subjects, suspicion of pregnancy
* Subject has received treatment with another investigational drug or device within the past 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
To determine the success rate in reaching within working distance of the Cecum with no complications. | 1 month

SECONDARY OUTCOMES:
To assess the ability to perform routine therapeutic interventions such as biopsies, polypectomies, APC etc. as compared to therapeutic interventions with standard colonoscopes found in the literature. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ori Segol, Dr., Principal Investigator — Carmel Medical Center